CLINICAL TRIAL: NCT05900817
Title: Esthetic Management of Anterior Teeth Utilizing Two Micro Abrasion Treatments: Randomized Clinical Trial
Brief Title: Esthetic Management of Anterior Teeth Utilizing Two Micro Abrasion Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Shafik Khalil, lecturer of Pediatric Dentistry and Dental public health, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #REC-FDBSU/06102020-01/SS
Record Dates: First submitted 2022-11-16; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hypomineralization of Enamel
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants, outcome assessors and data analyst will be blinded to the interventions during the clinical trial. After complete data entry of the trial, they will be unblinded to avoid any bias to either two groups. Outcome assessor chart was examined and filled up by two experts. Two principal Investigators and operators) will be blinded until generation of the allocation sequence. Later on, two invistigators will be unblinded within the treatment session due to different treatments packing and steps. Both investigators won't be involved in assessing the outcome. Informed Consent: both Investigators will be introduced the trial to patients regarding the main aspects of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- antivet arm (Experimental): Teeth treated will be isolated first then Vaseline will be placed on gingival sulcus before placing dental dam., patient will be seated at a 45 degree angle. Five drops of Antivet in the plastic mixing well that comes. Then ANTIVET solution will be applied over the tooth's surface using a well condensed cotton pellet (approximately a 3 mm diameter). When the cotton pellet is pigmented by the tooth's staining, it will be changed for a new one. This process may take about 1 to 5 minutes per tooth, It should take no longer than 15 minutes from the moment the solution contacts the tooth's surface
  Interventions: Other: antivet
- opulsture arm (Active Comparator): They were isolated with a rubber dam and then a fine-grit, water-cooled diamond bur was applied to the stained and white opaque enamel region for five to 10 seconds to enable penetration of the gel into the enamel. An approximately 1-mm- thick layer of 6.6% hydrochloric acid slurry with silicone carbide microparticles (Opalustre, Ultradent Products Inc, South Jordan, UT, USA) was applied to the affected tooth surfaces.
  Interventions: Other: Oplsture

INTERVENTIONS:
Other: antivet — A material used for micro abrasion of teeth
  Arms: antivet arm
Other: Oplsture — A material used for micro abrasion of teeth
  Arms: opulsture arm

SUMMARY:
the aim of this clinical trial is to compare the new micro-abrasion material "ANTIVET" compared to the conventional micro-abrasion material used widely "opalustre". to achieve better esthetics in cases of hypo-mineralized anterior permanent teeth of children and young adults.

both materials will be applied by the researchers and patient's teeth sensitivity and color change will be assessed immediately , after one month and after three months

DETAILED DESCRIPTION:
Materials and methods:

Enamel Microabrasion Even though only maxillary and mandibular hypominerlized incisors and canines were included in the current study, all teeth visible during smiling, laughing, or speaking were treated in this trial. The teeth were cleaned with pumice before treatment. Initial photographs of the teeth were taken.

Opalustre:

They were isolated with a rubber dam and then a fine-grit, water-cooled diamond bur was applied to the stained and white opaque enamel region for five to 10 seconds to enable penetration of the gel into the enamel. An approximately 1-mm- thick layer of 6.6% hydrochloric acid slurry with silicone carbide microparticles (Opalustre, Ultradent Products Inc, South Jordan, UT, USA) was applied to the affected tooth surfaces.

Antivet :

Teeth treated will be isolated first then Vaseline will be placed on gingival sulcus before placing dental dam., patient will be seated at a 45 degree angle. Five drops of Antivet in the plastic mixing well that comes. Then ANTIVET solution will be applied over the tooth's surface using a well condensed cotton pellet (approximately a 3 mm diameter). When the cotton pellet is pigmented by the tooth's staining, it will be changed for a new one. This process may take about 1 to 5 minutes per tooth, It should take no longer than 15 minutes from the moment the solution contacts the tooth's surface

Materials Treatment 1 opalustre Ultra dent Treatment 2 Antivet MDC

Sampling:

Thirty participants, aged between 9-18yrs, with dental hypo mineralized discolored anterior teeth and who met the following inclusion and exclusion criteria will be selected for the study.

Recruitment:

The two principal investigators and operators screened patients in Outpatient clinics of departments of Pediatric Dentistry and Public Health in Faculty of Dentistry - Beni-suef University & Restorative Dentistry- Faculty of Dentistry in the British University in Egypt irrespectively. The screening process was continued until the target population was achieved.

Patients will be randomly allocated in both treatment groups

Blinding:

Participants, outcome assessors and data analyst will be blinded to the interventions during the clinical trial. After complete data entry of the trial, they will be unblinded to avoid any bias to either two groups.

Outcome assessor chart was examined and filled up by two experts. Both investigators won't be involved in assessing the outcome. Informed Consent: both Investigators will be introduced the trial to patients regarding the main aspects of the trial.

A written informed consent forms (Arabic and English versions) were signed by all patients participated in the trial. The protocol, informed consent forms, participant education and recruitment materials will be reviewed and approved by the Ethical Committee of Faculty of Oral and Dental Medicine- Beni-Suef University.

outcomes will be assessed immediately after the procedure, 1 month and 3 months Pre-operative and post operative photographs will be taken to document color improvement in each visit

ELIGIBILITY:
Inclusion Criteria:

participants having anterior teeth

1. with Degree 1 (mild) according to the Wetzel and Reckel scale.: Isolated white and cream to yellowish brown discolorations on the chewing surface and upper part of the crown , for
2. caries-free teeth.

Exclusion Criteria:

were children with :

1. generalized hypoplasia
2. amelogenesis imperfecta
3. dentinogenesis imperfecta
4. tetracycline or diffuse hypoplasia like fluorosis
5. grossly broken and missing teeth where the reason of MIH could not be established.
6. children with special health care needs.
7. fractured, carious, grossly decayed teeth. -

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
postoperative changes in teeth sensitivity | change from baseline teeth sensitivity immediately after treatment ,change from baseline teeth sensitivity after one month from treatment and change from baseline teeth sensitivity after three month from treatment after
  visual analogue scale (0:no pain,10:worst pain) - verbal analogue scale (no pain or distressing, miserable pain )
patient satisfaction | after 3 months
  using a 5- point Likert scale ( 1= not at all satisfied, 5= extremely satisfied) likert scale: where 1 represents no improvement at all and 7 represents excellent improvement.
  photography conditions will be standardized during pre and post treatment photos

CONTACTS AND LOCATIONS:
Overall Officials: Sarah MS khalil, phD, Principal Investigator — lecturer of Pediatric Dentistry ,Faculty of Dentistry ,Beni-Suef University
Locations (1):
- Sarah Mohamed Shafik Khalil, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No
all Data will be available within 3 months

REFERENCES:
- [Background] Denis M, Atlan A, Vennat E, Tirlet G, Attal JP. White defects on enamel: diagnosis and anatomopathology: two essential factors for proper treatment (part 1). Int Orthod. 2013 Jun;11(2):139-65. doi: 10.1016/j.ortho.2013.02.014. Epub 2013 Apr 16. English, French. PMID 23597715
- [Background] Torres CR, Borges AB. Color masking of developmental enamel defects: a case series. Oper Dent. 2015 Jan-Feb;40(1):25-33. doi: 10.2341/13-346-T. Epub 2014 Aug 19. PMID 25136905
- [Background] Akin M, Basciftci FA. Can white spot lesions be treated effectively? Angle Orthod. 2012 Sep;82(5):770-5. doi: 10.2319/090711.578.1. Epub 2012 Feb 23. PMID 22356705
- [Background] Huang GJ, Roloff-Chiang B, Mills BE, Shalchi S, Spiekerman C, Korpak AM, Starrett JL, Greenlee GM, Drangsholt RJ, Matunas JC. Effectiveness of MI Paste Plus and PreviDent fluoride varnish for treatment of white spot lesions: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Jan;143(1):31-41. doi: 10.1016/j.ajodo.2012.09.007. PMID 23273358
- [Background] Pini NI, Sundfeld-Neto D, Aguiar FH, Sundfeld RH, Martins LR, Lovadino JR, Lima DA. Enamel microabrasion: An overview of clinical and scientific considerations. World J Clin Cases. 2015 Jan 16;3(1):34-41. doi: 10.12998/wjcc.v3.i1.34. PMID 25610848
- [Background] Deshpande AN, Joshi NH, Pradhan NR, Raol RY. Microabrasion-remineralization (MAb-Re): An innovative approach for dental fluorosis. J Indian Soc Pedod Prev Dent. 2017 Oct-Dec;35(4):384-387. doi: 10.4103/JISPPD.JISPPD_216_16. PMID 28914255
- [Background] Donly KJ, O'Neill M, Croll TP. Enamel microabrasion: a microscopic evaluation of the "abrosion effect". Quintessence Int. 1992 Mar;23(3):175-9. PMID 1641458